CLINICAL TRIAL: NCT03819023
Title: Validation of RespiLife for Detection of Respiratory Suppression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioresp Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BR01
Record Dates: First submitted 2019-01-15; First posted 2019-01-28 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Respiration Disorders
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Intervention Model Description: Evaluation of the device on people with normal and suppressed respiration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Normal subjects (No Intervention)
- respiratory suppressing drugs (Active Comparator)
  Interventions: Diagnostic Test: Respilife monitor

INTERVENTIONS:
Diagnostic Test: Respilife monitor — Respilife monitor
  Arms: respiratory suppressing drugs

SUMMARY:
The purpose of this study is to evaluate the accuracy of RespiLife diagnostic technology for detection of respiratory rate and oxygen saturation in human subjects. This includes evaluation of Bioresp's RespiLife and its accuracy for measurement of respiratory rate and oxygen saturation.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the accuracy of RespiLife diagnostic technology for detection of respiratory rate and oxygen saturation in human subjects. This includes evaluation of Bioresp's RespiLife and its accuracy for measurement of respiratory rate and oxygen saturation.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign the informed consent
* English speaking.
* Able to comply with visits and follow ups included in this protocol
* Ages 18-80 years

Exclusion Criteria:

* Mentally or cognitively incompetent persons who cannot understand the procedures or consent to the procedures.
* An unstable medical condition, acute of chronic, that in the opinion of the investigator puts the subject at health risks related this trial or interferes with the clinical trial and data collection.
* If a subject is not able to stop his CPAP or BiPAP therapy at least one week prior to the sleep study night. This will be determined ty the principal investigator based on her judgment.
* Skin rash on the forehead.
* A history of skin allergy to medical tape, even hypoallergenic tape.
* A history of skin cancer on the forehead.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-03-02 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
oxygen saturation percentage using photoplethysmography | 6 hours
  The Respilife algorithm will calculate the respiratory rate and oxygen saturation. The measurements will be compared and analyzed against the gold standard measurements using FDA -approved clinical tools, such as Nellcor oximeter and photoplethysmographer.
Respiratory rate, breaths per minute using photoplethysmography | 6 hours
  The Respilife algorithm will calculate the respiratory rate and oxygen saturation. The measurements will be compared and analyzed against the gold standard measurements using FDA -approved clinical tools, such as Nellcor oximeter and photoplethysmographer and piezo electric and respiratory inductance plethysmography.

CONTACTS AND LOCATIONS:
Locations (1):
- Peninsula Sleep Center, Burlingame, California, United States

IPD SHARING:
Plan to Share IPD: Undecided